CLINICAL TRIAL: NCT05959265
Title: Effect of Exercise Therapy on Psychological State and Clinical Prognosis of Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAMDD-001
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Lung Cancer
Keywords: Exercise; psychological; clinical prognosis; advanced non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1 (Experimental): Patients in the treatment group will undergo a 12-week intervention consisting of three 30-minute walking exercises per week during their standard cancer treatment. A personalized walking plan using fitness trackers will be provided to record each patient's daily average heart rate, step count, and additional steps and heart rate during the three 30-minute walking exercises per week to assess their activity levels. Weekly collaborations between the principal investigator and each participant will be conducted to assess step-related parameters.
  Interventions: Behavioral: exercise
- Arm2 (No Intervention): Patients in the control group will receive standard cancer treatment and will not be instructed to avoid exercise. They will also be provided with fitness trackers to record their daily average heart rate and step count to evaluate their daily activity level. Furthermore, participants will be retrospectively asked about their physical activity during the intervention period at the end of the intervention phase.

INTERVENTIONS:
Behavioral: exercise — Patients in the treatment group will undergo a 12-week intervention consisting of three 30-minute walking exercises per week during their standard cancer treatment. A personalized walking plan using fitness trackers will be provided to record each patient's daily average heart rate, step count, and additional steps and heart rate during the three 30-minute walking exercises per week to assess their activity levels. Weekly collaborations between the principal investigator and each participant will be conducted to assess step-related parameters.
  Arms: Arm1

SUMMARY:
This study is an open-label, prospective, two-arm clinical trial aimed at evaluating the impact of exercise therapy on the psychological state and clinical prognosis of advanced non-small cell lung cancer (NSCLC) patients.

After signing the informed consent form, patients will be randomly assigned to either the treatment group or the control group. Enrolled patients will undergo both a treatment phase and a follow-up phase. Patients in the treatment group will undergo a 12-week intervention consisting of three 30-minute walking exercises per week during their standard cancer treatment. A personalized walking plan using fitness trackers will be provided to record each patient's daily average heart rate, step count, and additional steps and heart rate during the three 30-minute walking exercises per week to assess their activity levels. Weekly collaborations between the principal investigator and each participant will be conducted to assess step-related parameters.Additionally, the primary investigator of the study will conduct two investigator-led structured counseling sessions at the beginning of the project and midway through the intervention. These sessions will include a comprehensive assessment of the participant's lifestyle and current symptoms. Recommendations and counseling, such as symptom management, will be provided immediately following the investigator-led sessions and continuously throughout the study, along with appropriate referrals or contacts.Patients in the control group will receive standard cancer treatment and will not be instructed to avoid exercise. They will also be provided with fitness trackers to record their daily average heart rate and step count to evaluate their daily activity level. Furthermore, participants will be retrospectively asked about their physical activity during the intervention period at the end of the intervention phase.During the follow-up phase, researchers will provide appropriate treatment advice based on the patients' conditions. Completed study patients will undergo follow-up assessments every three months for one year.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Pathologically confirmed IIIB/IV stage NSCLC patients;
3. According to the judgment of the researcher, it is suitable for enrollment;
4. Can walk independently without assistance;
5. The subjects voluntarily joined this study and signed an informed consent form, with good compliance and cooperation in follow-up.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Severe active infection
3. Unable to walk
4. Cannot be active (more than two days)
5. Severe neurological or cardiac damage
6. Severe respiratory insufficiency
7. Uncontrollable pain
8. Those who have perceptual barriers or cognitive and Communication disorder and are unable to cooperate;
9. Participated in other sports groups during the research period;
10. According to the judgment of the researchers, the subjects may have other factors that may lead to the forced termination of this study, such as other serious illnesses (including mental illness) requiring concurrent treatment, serious laboratory test abnormalities, accompanied by family or social factors, which may affect the safety of the subjects, or the collection of data and samples;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 3 months
  Changes in anxiety scores measured through the Hospital Anxiety and Depression Scale
ORR (Objective Response Rate) | 3 months
  ORR (Objective Response Rate) is defined as the proportion of participants who confirmed at least one CR (Complete Response) or PR (Partial response) before disease progression based on Response Evaluation Criteria in Solid Tumors (RECIST)1.1 as assessed by the investigator.

SECONDARY OUTCOMES:
Depression | 3 months
  Changes in depression scores measured through the Hospital Anxiety and Depression Scale
Tumor biomarker | 3 months
  NSE、CEA、CA125、CA153、CYFRA21-1、SCC
adiponectin | 3 months
  It is an endogenous bioactive peptide or protein secreted by adipocytes
Inflammatory biomarker | 3 months
  PCT、CRP、TNF、IL-6、IL-8 和 IL-2, IL-13, IL-18
OS (Overall Survival) | 1 year
  OS (Overall Survival) is defined as the time from the initial administration of treatment to the date of death due to any cause. Patients who have not died at the time of statistical analysis will have their survival time censored at the last known date of their survival.
PFS (Progression-Free Survival) | 1 year
  PFS (Progression-Free Survival) is defined as the time between the onset of randomization and the occurrence (progression) or death (for any reason) of the tumor

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University